CLINICAL TRIAL: NCT01009996
Title: Kissing Drug-Eluting Balloons After Bare Metal Stenting of Coronary Bifurcation Lesions.
Brief Title: Efficacy Study of Kissing Drug-Eluting Balloons in Coronary Bifurcation Lesions
Acronym: KISSING DEBBIE
Status: Withdrawn | Type: Observational
Why Stopped: Funding issues
Sponsor: Ospedale Santa Maria Goretti (Other)
Responsible Party: Principal Investigator, Gregory Sgueglia, MD, Principal investigator, Ospedale Santa Maria Goretti
Other Study IDs: SMG-003
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Coronary Artery Disease; Bifurcation Lesions
Keywords: Coronary bifurcation lesions
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Coronary bifurcation lesions
  Interventions: Procedure: Kissing DEB

INTERVENTIONS:
Procedure: Kissing DEB — Provisional bare metal stenting followed by kissing drug-eluting balloons

SUMMARY:
KISSING DEBBIE's aim at assessing angiographic and clinical outcomes of provisional treatment of coronary bifurca6on lesions according to TAP sten6ng with BMS and final kissing DEB

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* De novo major bifurca6on lesion of the left coronary artery (LAD-D; LCX-OM)
* RVD 2.25-4.0 mm

Exclusion Criteria:

* LMCA
* AMI within 48 hours
* Limited compliance with 3-month dual antiplatelet therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All coming
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-10 (Estimated); Primary Completion 2011-02 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Late lumen loss on both MV and SB | 9 months

SECONDARY OUTCOMES:
Procedural success (residual stenosis <20% on MV and <50% on SB with TIMI flow 3 for both) | immediate
Binary restenosis rate | 9 months
Major adverse cardiac events | 3 months
Major adverse cardiac events | 6 months
Major adverse cardiac events | 9 months
Major adverse cardiac events | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- UOC Emodinamica e Cardiologia Interventistica - Ospedale Santa Maria Goretti, Latina, Italy

REFERENCES:
- [Derived] Sgueglia GA, Todaro D, Bisciglia A, Conte M, Stipo A, Pucci E. Kissing inflation is feasible with all second-generation drug-eluting balloons. Cardiovasc Revasc Med. 2011 Sep-Oct;12(5):280-5. doi: 10.1016/j.carrev.2010.12.001. Epub 2011 Jan 26. PMID 21273144